CLINICAL TRIAL: NCT03394534
Title: 'Comprehensive Geriatric Assessment' for Older Adults With Frailty Within Primary Care Setting: A Randomised Feasibility Trial
Brief Title: Comprehensive Geriatric Assessment in Primary Care: A Randomised Feasibility Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Derby (Other)
Collaborators: Derbyshire Clinical Commissioning Groups (Unknown)
Responsible Party: Principal Investigator, Reza Safari, Research Fellow, University of Derby
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: v3.6
Record Dates: First submitted 2017-12-18; First posted 2018-01-09 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Frailty
Keywords: Comprehensive Geriatric Assessment; Frailty; electronic Frailty Index; eFI; Care and Support plan; Primary Care
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CGA group (Experimental)
  Interventions: Other: CGA group
- Treatment as Usual (No Intervention)

INTERVENTIONS:
Other: CGA group — CGA Plus Individualised Care and Support Plan delivered by Advanced Clinical Practitioner (ACP)
  Arms: CGA group

SUMMARY:
The study aims to explore feasibility of implementing a tailored CGA to older adults with frailty and evaluate staff and patients perception of the intervention. In line with this, the objectives of the study are:

1. To assess applicability of finding older adults with frailty using eFI and delivering subsequent CGA and care planning at patients' home
2. To investigate staff and older adults' perception of CGA programme
3. To assess the health care resource usage and cost of the CGA programme
4. To measure key health related outcome domains including function, quality of life, loneliness, pain, falls and mobility.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 to 95 years
* eFI score > 0.12

Exclusion Criteria:

* Do not meet criteria for frailty based on Gait speed, timed up and go test and PRISMA questionnaire

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-06-15 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Hospitalisation and Nursing Home Admissions | at 6 months post intervention
  Number of hospital and/or care home admissions during the 6 months period and reported in terms of admitted v. not admitted

SECONDARY OUTCOMES:
Functional Status | at baseline and 6 months post intervention
  Improve Patient functional ability measured using Functional Independence Measure (FIM) questionnaire total score
Loneliness | at baseline and 6 months post intervention
  Improve overall, emotional, and social loneliness calculated using the De Jong Gierveld Loneliness Scale total score. The scale is used to assess subjective perception of social participation or isolation in elderly adults.
Health related Quality of Life | at baseline and 6 months post intervention
  Change in health related quality of life calculated using the 36-Item Short Form Survey (SF-36). The Sf-36 is patient reported outcome measure with a set of generic quality of life measures including vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, mental health subscales.
Number of 999 calls and A+E attendance during the 6 months period | at 6 months post intervention
Length of time spent on A+E during the 6 months period | at 6 months post intervention
Length of time stayed in hospital or care home during the 6 months period | at 6 months post intervention
Therapist and staff time spent on CGA during the 6 months period | at 6 months post intervention
Number of GP/GP out of office attendance (including calls to GP) during the 6 months period | at 6 months post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Reza Safari, PhD, Principal Investigator — University of Derby
Locations (1):
- University of Derby, Derby, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Edmans J, Bradshaw L, Gladman JR, Franklin M, Berdunov V, Elliott R, Conroy SP. The Identification of Seniors at Risk (ISAR) score to predict clinical outcomes and health service costs in older people discharged from UK acute medical units. Age Ageing. 2013 Nov;42(6):747-53. doi: 10.1093/ageing/aft054. Epub 2013 May 10. PMID 23666405
- [Background] Clegg A, Young J, Iliffe S, Rikkert MO, Rockwood K. Frailty in elderly people. Lancet. 2013 Mar 2;381(9868):752-62. doi: 10.1016/S0140-6736(12)62167-9. Epub 2013 Feb 8. PMID 23395245
- [Background] Gladman JR, Conroy SP, Ranhoff AH, Gordon AL. New horizons in the implementation and research of comprehensive geriatric assessment: knowing, doing and the 'know-do' gap. Age Ageing. 2016 Mar;45(2):194-200. doi: 10.1093/ageing/afw012. PMID 26941353
- [Background] Fit for Frailty - Developing, commissioning and managing services for people living with frailty in community settings - a report from the British Geriatrics Society and the Royal College of General Practitioners 2015.
- [Background] Clegg A, Rogers L, Young J. Diagnostic test accuracy of simple instruments for identifying frailty in community-dwelling older people: a systematic review. Age Ageing. 2015 Jan;44(1):148-52. doi: 10.1093/ageing/afu157. Epub 2014 Oct 29. PMID 25355618
- [Derived] Safari R, Jackson J, Boole L. Comprehensive geriatric assessment delivered by advanced nursing practitioners within primary care setting: a mixed-methods pilot feasibility randomised controlled trial. BMC Geriatr. 2023 Aug 24;23(1):513. doi: 10.1186/s12877-023-04218-0. PMID 37620760